CLINICAL TRIAL: NCT04380051
Title: Evaluation of a Sensory-tonic Stimulation on Development of Parent-infant Interaction and Social Cognition in Very Premature Children
Brief Title: Evaluation of a Sensory-tonic Stimulation on Development of Parent-infant Interactions and Social Cognition in Very Premature Children
Acronym: CALIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR20064*
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Very Preterm Birth

STUDY DESIGN:
Intervention Model Description: participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 : skin-to-skin contact associated with a sensory-tonic s (Experimental): skin-to-skin contact left free for parents associated with a sensory-tonic stimulation five times a week during 15 minutes at each time
  Interventions: Behavioral: sensory-tonic stimulation; Behavioral: skin-to-skin contact
- Arm 2 : skin-to-skin contact only (Active Comparator): skin-to-skin contact left free for parents
  Interventions: Behavioral: skin-to-skin contact

INTERVENTIONS:
Behavioral: sensory-tonic stimulation — sensory-tonic stimulation done by the parents to the child, five times a week during 15 minutes at each time
  Arms: Arm 1 : skin-to-skin contact associated with a sensory-tonic s
Behavioral: skin-to-skin contact — skin-to-skin contact left free for parents

SUMMARY:
Attachment is built primarily on the first interactions of the first 9 months of a baby's life. These first interactions and their effects of stress, pleasure and displeasure are retained to establish some of the baby's attachment behaviours and future relationships with others.

Extreme prematurity strongly modify these first interactions between parents and child. Very preterm child is separated from his parents and is placed in a stressful, technical and potentially painful environment.

Early interventions stimulate neuroplasticity and can positively affect the neurological development of very preterm infant. Tactile stimuli such as skin-to-skin contact and massages carried out by parents can be pleasant experiences that can support early interactions between parents and child.

DETAILED DESCRIPTION:
The aim of the study is to evaluate impact of a sensory-tonic stimulation on development of parent-infant interaction and on social cognition in very premature children.

ELIGIBILITY:
inclusion criteria :

* very preterm child (born before 32 weeks of amenorrhoea)
* parents agreeing to participate to the study

exclusion criteria :

* child born before 25 weeks of amenorrhoea
* child with a birth weight less than 600 grams
* child with congenital malformation
* child with hemodynamic instability

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2027-01-19 (Estimated); Study Completion 2033-01-19 (Estimated)

PRIMARY OUTCOMES:
interactions between parents and child | 12 months
  Two free play sequences of 15 minutes will be filmed. The Coding Interactive Behavior (CIB; Feldman, 1998) contains 43 items (22 relating to parents, 16 relating to child and 5 related to parent-child dyad. Each item is rated from 1 (a little) to 5 (a lot). The Coding Interactive Behavior has 6 dimensions. The dimension "social commitment of the child" will be the primary outcome for this study.

SECONDARY OUTCOMES:
Social cognition / Theory of mind | 6 years
  small stories involving the thinking and feelings of character

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guittard C, Novo A, Eutrope J, Gower C, Barbe C, Bednarek N, Rolland AC, Caillies S, Loron G. Protocol for a prospective multicenter longitudinal randomized controlled trial (CALIN) of sensory-tonic stimulation to foster parent child interactions and social cognition in very premature infants. Front Pediatr. 2023 Jan 16;10:913396. doi: 10.3389/fped.2022.913396. eCollection 2022. PMID 36727004